CLINICAL TRIAL: NCT05878431
Title: The Effect of Foot Reflexology Applied on Diabetic Patients With Neuropathic Pain on the Patients' Quality of Life, Hope and Pain Levels
Brief Title: Foot Reflexology in Diabetic Patients With Neuropathic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Principal Investigator, Cihat Demirel, Lecturer, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Reflexology
Record Dates: First submitted 2023-03-27; First posted 2023-05-26 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus; Patient Engagement; Reflexology
Keywords: Reflexology; Diabetes Mellitus; Neuropathic Pain; Hope; Quality of Life
MeSH Terms: conditions — Diabetes Mellitus; Patient Participation; Neuralgia

STUDY DESIGN:
Intervention Model Description: This study was conducted as a single-blind randomized controlled study with pretest-posttest
Who Masked: Participant
Masking Description: In this study, patients were randomized to the experimental and control groups by using a simple random numbers table from the computer-assisted randomization program in accordance with the simple random sampling method. In this study, participants in the experimental and control groups were blind to each other; however, the researcher was not blinded to the group allocation as he was also the practitioner.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental groups (Experimental): patients in the experimental group during the pre-test phase; "Patient Information Form", "Herth Hope Scale", "Four-Question Neuropathic Pain Questionnaire (DN4Q)", "The Effect of Neuropathic Pain on Quality of Life Questionnaire (NePIQOL)" and "Visual Analog Scale (VAS)" were administered by face-to-face interview technique. Then to the patients in the experimental group; A total of 12 sessions of foot reflexology, two sessions per week, were applied for 6 weeks. patients in the experimental group during the pos-test phase; "Herth Hope Scale", "Four-Question Neuropathic Pain Questionnaire (DN4Q)", "The Effect of Neuropathic Pain on Quality of Life Questionnaire (NePIQOL)" and "Visual Analog Scale (VAS)" were administered by face-to-face interview technique
  Interventions: Other: Foot Reflexology
- Control groups (No Intervention): patients in the control group at the pre-test stage; "Patient Information Form", "Herth Hope Scale", "Four-Question Neuropathic Pain Questionnaire (DN4Q)", "The Effect of Neuropathic Pain on Quality of Life Questionnaire (NePIQOL)" and "Visual Analog Scale (VAS)" were applied. with face-to-face interview technique. patients in the control group during the pos-test phase; "Herth Hope Scale", "Four-Question Neuropathic Pain Questionnaire (DN4Q)", "The Effect of Neuropathic Pain on Quality of Life Questionnaire (NePIQOL)" and "Visual Analog Scale (VAS)" were administered by face-to-face interview technique

INTERVENTIONS:
Other: Foot Reflexology — The patients in the experimental group underwent 12 sessions of foot reflexology in a quiet room, twice a week, for 6 weeks. No application was made to the patients in the control group.
  FOOT REFLEXOLOGY APPLICATION STAGES
  * Application of heating methods such as Achilles tendon stretching, wrist loosening, walking the thumbs of both hands on the soles of the feet and wringing the laundry, which lasts about 3 minutes,
  * Pressure on the brain, cervical region, solar plexus (the projection of the central nervous system on the sole of the foot), lymph system, adrenal glands, urinary system, digestive system, sciatic nerve, hips, knees and reflex points on the soles of the legs for about 10-15 minutes. implementation (Figure 3.4),
  * Ending the application by applying heating methods such as Achilles tendon stretching, wrist loosening, walking the thumbs of both hands on the soles of the feet and wringing the laundry, which lasts approximately 3 minutes after the application.
  Arms: Experimental groups

SUMMARY:
This study was carried out to determine the effect of foot reflexology applied to diabetic patients with neuropathic pain on their quality of life, hope and pain levels.

This research, which was designed as a randomized controlled and experimental study, was conducted between January 2022 and December 2022. It was determined that foot reflexology application increased the quality of life and hope level of diabetic patients with neuropathic pain and decreased the level of pain.

DETAILED DESCRIPTION:
Aim: This study was carried out to determine the effect of foot reflexology applied to diabetic patients with neuropathic pain on their quality of life, hope and pain levels.

Material and Method: This research, which was designed as a randomized controlled and experimental study, was conducted between January 2022 and December 2022. The data of the study consisted of 102 diabetic patients with neuropathic pain, 51 of whom were experimental and 51 were controls. As data collection tools; Patient Information Form, Herth Hope Scale (HHI), Four-Question Neuropathic Pain Questionnaire (DN4Q), Neuropathic Pain Impact on Quality of Life Questionnaire (NePIQoL), and Visual Analog Scale (VAS) were used. A total of 12 sessions of foot reflexology were applied to the patients in the experimental group, twice a week for 6 weeks. No intervention was performed on the patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Do not have any physical or mental illness that will prevent communication,
* Diabetic neuropathic pain [with a total score of at least 4 and above according to the Four-Question Neuropathic Pain Questionnaire (DN4Q)]
* Patients who can read, write and speak Turkish

Exclusion Criteria:

* Complications developing during reflexology practice,
* Not attending at least one of the practice sessions,
* It was planned to exclude patients who wanted to leave at any stage of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Vizüel Analog Scale (VAS) | At the end of the 6-week intervention
Herth Hope Scale | At the end of the 6-week intervention
Neuropathic Pain Impact on Quality of Life Questionnaire (NePIQOL) | At the end of the 6-week intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Mus State Hospital, Muş, Muş, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No